CLINICAL TRIAL: NCT04290468
Title: Role of Ultrasound in Shoulder Impingement
Brief Title: Dynamic Ultrasound in Shoulder Impingement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Ismail Ahmed Mohammed, principal investigator, Assiut University
Other Study IDs: ultrasound in shoulder
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dynamic ultrasound — The ultrasound examination will be carried out blinded to the results of MRI using the Affiniti 70 ultrasound machine by Philips (USA) via a 5-12MHz linear transducer.
  MRI was performed on a high field system (1.5 Tesla) magnet units (Philips Acheiva).
  Other Names: MRI

SUMMARY:
* To evaluate the role of dynamic ultrasound in evaluation patient with clinically suspected shoulder joint impingement.
* To assess the added value of dynamic ultrasonography to the static examination of patients with clinically suspected impingement.

DETAILED DESCRIPTION:
Shoulder impingement syndromes and degenerative rotator cuff (RC) disease represent the main causes of shoulder pain . Impingement is classified into four types, depending on the site of soft-tissue entrapment: sub acromial, sub coracoid, poster superior inner and anterosuperior inner impingement. The sub acromial impingement syndrome is by far the most common in practice. . The clinical symptoms of sub acromial impingement include nocturnal pain and progressive, limited range of motion. At clinical examination, there is a painful area at 80-120° elevation, which is worsened during downward movements Osteophytes, or an abnormal shape of the acromion, sub acromial spurs, and the acromioclavicular joint, are common causes of compression at the rotator cuff and the overlying subacromial-subdeltoid bursa . Ultrasonography (US) is a commonly performed examination for shoulder impingement, recommended by experts as the first-choice technique to evaluate various shoulder diseases. Shoulder impingement is the most common and well-recognized indication for dynamic US in the shoulder.

Dynamic evaluation can be done by shoulder abduction or flexion with the probe placed at the end of the acromion in the coronal plane or in the sagittal plane. The two important points to be checked for shoulder impingement are the humeral head depression and tendon/bursal impingement . Because humeral head depression is essential to make enough space for the rotator cuff to slide beneath the acromion, the center of the humeral head normally moves inferiorly in the latter half of the cycle during shoulder abduction. When the humeral head does not move inferiorly or abnormally moves superiorly, the space for the rotator cuffs and the subacromial-subdeltoid bursa decreases and subacromial impingement can occur .

Magnetic resonance imaging (MRI) is currently considered the reference standard for imaging of shoulder disorders. The strength of MRI lies in its ability to assess sonographically inaccessible areas such as labrum, deep parts of various ligaments, capsule, and areas obscured by bone . MRI is the imaging study of choice for classifying tendon retraction and assessing the shoulder musculature. Its main disadvantage is being a static evaluation of the shoulder joint . There are several advantages of Ultrasonography over MRI. Ultrasonography has the benefit of being a dynamic form of imaging as compared to the static MRI. Ultrasonography is portable, quick, and a more cost-effective method. It is also better tolerated by the patient and allows interaction with the patient, who can point at the symptomatic area, thus optimizing the diagnostic yield.

ELIGIBILITY:
Inclusion Criteria

* All patients referred to the Radiology department with clinically suspected shoulder impingement. Inclusion Criteria:

Exclusion Criteria:

* The following categories of patient will be excluded from the study.

  1. History of previous shoulder surgery.
  2. History of joint dislocation.
  3. Fracture to the shoulder girdle.
  4. Patient with contraindication to MRI.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: sample size was determined by using G*power version 3.1.9.2 for windows for power analysis .we estimated 37 patients to be included in the study with statistically power 95% and 0.05 as an alpha error
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
comparison of dynamic ultrasound findings with MRI | Baseline
  To determine the role of dynamic shoulder ultrasound in evaluation of patients with clinically suspected shoulder impingement

REFERENCES:
- [Background] Rowbotham EL, Grainger AJ. VIDEO: Ultrasound Evaluation of External Shoulder Impingement. AJR Am J Roentgenol. 2018 Aug;211(2):W122. doi: 10.2214/AJR.18.19534. Epub 2018 Jun 21. PMID 29927333
- [Background] Coats-Thomas MS, Massimini DF, Warner JJP, Seitz AL. In Vivo Evaluation of Subacromial and Internal Impingement Risk in Asymptomatic Individuals. Am J Phys Med Rehabil. 2018 Sep;97(9):659-665. doi: 10.1097/PHM.0000000000000940. PMID 29613881
- [Background] Pesquer L, Borghol S, Meyer P, Ropars M, Dallaudiere B, Abadie P. Multimodality imaging of subacromial impingement syndrome. Skeletal Radiol. 2018 Jul;47(7):923-937. doi: 10.1007/s00256-018-2875-y. Epub 2018 Feb 14. PMID 29445933
- [Background] Soker G, Gulek B, Soker E, Kaya O, Inan I, Arslan M, Esen K, Memis D, Yilmaz C. Sonographic assessment of subacromial bursa distension during arm abduction: establishing a threshold value in the diagnosis of subacromial impingement syndrome. J Med Ultrason (2001). 2018 Apr;45(2):287-294. doi: 10.1007/s10396-017-0839-9. Epub 2017 Oct 26. PMID 29075914
- [Background] Do HK, Lim JY. Ultrasonographic Evaluation and Feasibility of Posterosuperior Internal Impingement Syndrome: A Case Series. PM R. 2017 Jan;9(1):88-94. doi: 10.1016/j.pmrj.2016.06.008. Epub 2016 Jun 16. PMID 27317919
- [Background] Daghir AA, Sookur PA, Shah S, Watson M. Dynamic ultrasound of the subacromial-subdeltoid bursa in patients with shoulder impingement: a comparison with normal volunteers. Skeletal Radiol. 2012 Sep;41(9):1047-53. doi: 10.1007/s00256-011-1295-z. Epub 2011 Oct 14. PMID 21997670
- [Background] Michener LA, Subasi Yesilyaprak SS, Seitz AL, Timmons MK, Walsworth MK. Supraspinatus tendon and subacromial space parameters measured on ultrasonographic imaging in subacromial impingement syndrome. Knee Surg Sports Traumatol Arthrosc. 2015 Feb;23(2):363-9. doi: 10.1007/s00167-013-2542-8. Epub 2013 Jun 5. PMID 23736252